CLINICAL TRIAL: NCT06156020
Title: Analysis of Operative Outcomes Following Endoscopic Resection of Pituitary Adenomas
Brief Title: Outcome Analysis of Endoscopic Resection of Pituitary Adenomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-ER-112-452
Record Dates: First submitted 2023-11-15; First posted 2023-12-05 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-11

CONDITIONS: Pituitary Adenoma
Keywords: pituitary adenoma
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic endonasal surgery (Other): Patients who received endoscopic endonasal resection of pituitary adenomas
  Interventions: Procedure: Endoscopic endonasal surgery

INTERVENTIONS:
Procedure: Endoscopic endonasal surgery — Endoscopic endonasal transsphenoidal approach for resection of pituitary adenomas

SUMMARY:
The goal of this prospective study is to learn about the operative outcomes in patients with pituitary adenoma who receive endoscopic resection.

The main question it aims to answer is:

• What are the outcomes of patient following endoscopic resection? including visual, hormonal, survival, and functional outcomes.

Participants' data including clinical history, laboratory data, radiographic images, intraoperative videos will be evaluated and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Pathological diagnosis of pituitary adenoma
* Underwent endoscopic endonasal resection

Exclusion Criteria:

* Age < 18 or > 80 years
* Non-pituitary adenoma pathologies
* Underwent non-endoscopic surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Visual field | 6 months
  The postoperative visual field will be assessed with standard visual perimetry and compared with preoperative measurements.
Diabetes insipidus | 6 months
  Postoperatively, the patient's urine output and urine specific gravity will be measured to determine if the patient had diabetes insipidus. If the patient had diabetes insipidus, the duration of the diabetes insipidus will be recorded.
Cortisol level | 6 months
  Postoperative serum cortisol level will be measured and compared to preoperative levels.
Thyroid hormone level | 6 months
  Postoperative serum TSH and free T4 level will be measured and compared to preoperative levels.
Prolactin level | 6 months
  Postoperative serum prolactin level will be measured and compared to preoperative levels.
IGF-1 level | 6 months
  Postoperative serum IGF-1 level will be measured and compared to preoperative levels.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong CE, Chen PW, Hsu HJ, Cheng SY, Fan CC, Chen YC, Chiu YP, Lee JS, Liang SF. Collaborative Human-Computer Vision Operative Video Analysis Algorithm for Analyzing Surgical Fluency and Surgical Interruptions in Endonasal Endoscopic Pituitary Surgery: Cohort Study. J Med Internet Res. 2024 Jul 4;26:e56127. doi: 10.2196/56127. PMID 38963694